CLINICAL TRIAL: NCT02165345
Title: Long-Term Extension Study to Evaluate the Safety and Efficacy of Subcutaneous Tocilizumab in Patients With Polyarticular-Course and Systemic Juvenile Idiopathic Arthritis
Brief Title: Extension Study Evaluating the Safety and Efficacy of Subcutaneous Tocilizumab (RoActemra/Actemra) Administration in Systemic and Polyarticular-Course Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA29231; 2013-005212-98 (EudraCT Number)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental): Participants will receive tocilizumab until the commercial availability of the drug or up to 5 years, whichever is earlier.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — 162 mg tocilizumab will be administered by SC injection at the following intervals: pJIA participants less than (<) 30 kilograms (kg): every 3 weeks; pJIA participants greater than or equal to (>=) 30 kg: every 2 weeks; sJIA participants <30 kg: every 2 weeks; sJIA participants >/= 30 kg: once weekly
  Other Names: RoActemra, Actemra

SUMMARY:
This open-label extension of the JIGSAW studies (WA28117 [NCT01904279] and WA28118 [NCT01904292]) is designed to evaluate the long-term safety and efficacy of subcutaneous (SC) tocilizumab treatment in participants with polyarticular-course and systemic juvenile idiopathic arthritis (pJIA and sJIA). Participants from the 2 JIGSAW studies will continue to receive 162 milligrams (mg) of SC tocilizumab with treatment schedule according to arthritis subtype and body weight. Participants will receive the treatment until commercial availability of the drug or for a maximum of 5 years, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* Completion of either of the JIGSAW studies, study WA28117 (for participants with pJIA) or study WA28118 (for participants with sJIA)
* Adequate disease control with the use of SC tocilizumab(TCZ)(comparable to the use of IV TCZ, if received prior to enrollment in the JIGSAW study), per clinical judgment of the investigator
* For participants of reproductive potential: agreement to remain abstinent or use of effective contraception as defined by the study protocol

Exclusion Criteria:

* Prior discontinuation of SC tocilizumab because of inadequate clinical response during participation in a JIGSAW study
* Poorly controlled disease (in opinion of treating physician) despite treatment with SC tocilizumab in the JIGSAW study
* Prior discontinuation of intravenous tocilizumab because of inadequate clinical response or safety events (including hypersensitivity)
* Therapy with biologic agents (except tocilizumab) in the period between completion of the JIGSAW study and screening for the current study
* Concurrent treatment with disease-modifying anti-rheumatic drugs (DMARDs) (including methotrexate), nonsteroidal anti-inflammatory drugs (NSAIDs), and oral corticosteroids is permitted at the discretion of the investigator
* Use of live or attenuated vaccines and immunosuppressants, such as cyclosporine and cyclophosphamide
* Any significant concurrent medical or surgical conditions or findings that would jeopardize the participant's safety or ability to complete the study, including but not limited to disease of the nervous, renal, hepatic, cardiac, pulmonary, gastric, or endocrine system or any infection
* History of alcohol, drug, or chemical abuse within 6 months prior to screening
* History of atypical tuberculosis (TB) or active TB requiring treatment within 2 years prior to screening
* Known human immunodeficiency virus infection or other acquired forms of immune compromise or inborn conditions characterized by a compromised immune system
* Clinical signs or symptoms of acute or chronic viral hepatitis or chronic autoimmune hepatitis arising since enrollment in the JIGSAW study
* History of concurrent serious gastrointestinal disorders, such as ulcer or inflammatory bowel disease, Crohn's disease, ulcerative colitis, or other symptomatic lower gastrointestinal conditions
* History of or current cancer or lymphoma
* Uncontrolled diabetes mellitus with elevated glycosylated hemoglobin (HbA1c), defined with the use of age-specific standards
* Any abnormal laboratory values, an elevation of hepatic transaminases ([aspartate aminotransferase [AST] or alanine aminotransferase [ALT]), lowering of neutrophil count, or thrombocytopenia attributed to tocilizumab use by investigator at screening, the participant may be enrolled; however, the initial tocilizumab dose may be delayed to adhere to the protocol risk mitigation strategy or per the investigator's clinical judgment
* Prior stem cell transplant at any time

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Juvenile Arthritis Disease Activity Score (JADAS-71) | Baseline up to 3 years
Percentage of Participants With Adverse Events (AEs), Serious AEs (AEs) and AEs of Special Interest | Baseline up to 5 years

SECONDARY OUTCOMES:
Childhood Health Assessment Questionnaire (CHAQ) Score | Baseline up to 3 years
Percentage of Participants With Protocol Defined Inactive Disease/Clinical Remission | Baseline up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (9):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - University of Chicago Hospital, Chicago, Illinois
  - Hackensack University Medical Center; Pediatric Rheumatology, Hackensack, New Jersey
  - Duke University, Durham, North Carolina
  - Cincinnati Children'S Hospital Medical Center; Division of Rheumatology, Cincinnati, Ohio
  - Cleveland Clinic Fndn, Cleveland, Ohio
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - University of Utah; Immunology/Rheumatology/Allergy, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Argentina (2):
  - Hospital Gral de Niños Pedro Elizalde, Buenos Aires
  - Hospital de Ninos de la Santisima Trinidad; Hematología, Córdoba
- Australia (2):
  - Westmead Hospital; Paediatric Rheumatology, Westmead, New South Wales
  - Royal Children'S Hospital; Paediatric Rheumatology, Parkville, Victoria
- Brazil (2):
  - Universidade Federal de Sao Paulo - UNIFES, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Canada (2):
  - Alberta Children'S Hospital, Calgary, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
- CH de Bicêtre; Pediatrie Generale, Le Kremlin-Bicêtre, France
- Germany (3):
  - Charité Campus; Virchow Klinikum Berlin, Berlin
  - Uniklinikum Freiburg Zentrum für Kinder- und Jugendmedizin; Pädiatrische Infektio- u. Rheumatologie, Freiburg im Breisgau
  - Asklepios Klinik; Zentrum für Allgemeine Pädiatrie und Neonatologie, Sankt Augustin
- Irccs Ospedale Pediatrico Bambin Gesu - Dip. Di Medicina, Rome, Lazio, Italy
- Mexico (2):
  - Hospital Infantil de México "Federico Gomez"; Rheumatology, México
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez; Pediatria, Monterrey
- SI Sceintific children health center RAMS, Moscow, Russia
- Spain (4):
  - Hospital Sant Joan De Deu; Servicio de Reumatologia Pediatrica, Esplugas de Llobregat, Barcelona
  - Hospital Ramon y Cajal ; Servicio de Reumatologia, Madrid
  - Hospital de La Paz; Unidad de Reumatologia Pediatrica, Madrid
  - Hospital Universitario la Fe: Servicio de Reumatologia Pediatrica, Valencia
- United Kingdom (2):
  - Bristol Royal Hospital for Children; Rheumatology Department, Bristol
  - Alder Hey Children's NHS Foundation Trust, Liverpool

REFERENCES:
- [Derived] Brunner HI, Ruperto N, Ramanan AV, Horneff G, Minden K, Calvo Penades I, Alexeeva E, Cleary G, Stern SM, Kone-Paut I, Maldonado Velazquez MDR, Rabinovich CE, Remesal A, Silva CA, Nikishina I, Zucchetto M, Brockwell L, Gordon O, Nagel S, De Benedetti F; PRINTO and PRCSG Investigators. Long-term efficacy and safety of subcutaneous tocilizumab in clinical trials of polyarticular or systemic juvenile idiopathic arthritis. Rheumatology (Oxford). 2024 Sep 1;63(9):2535-2546. doi: 10.1093/rheumatology/keae180. PMID 38552315